CLINICAL TRIAL: NCT05361577
Title: Using a TENS System (Transcutaneous Electrical Noninvasive Stimulation) to Improve Pain Related to Fibromyalgia (EXOFIB)
Brief Title: Exopulse Mollii Suit and Fibromyalgia
Acronym: EXOFIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut De La Colonne Vertebrale Et Des Neurosciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-A01668-33
Record Dates: First submitted 2022-01-24; First posted 2022-05-04 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Fibromyalgia, Primary
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Phase 1: randomized sham controlled crossover study (active versus sham condition)
  Phase 2: Open label study (active condition)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active astimulation (Active Comparator): Active sessions will last 1 hour each. The following parameters will be used for electric stimulation: low frequency (20 Hz), low current intensity (2 mA), with a small pulse width of 25-170 microseconds.
  Interventions: Device: Exoplulse Mollii suit
- Sham stimulation (Sham Comparator): In the sham condition, the control unit will be programmed to start stimulating for 1 minute then it will shut off.
  Interventions: Device: Exopulse Mollii suit (sham)

INTERVENTIONS:
Device: Exoplulse Mollii suit — Exopulse Mollii suits consists of a body Garments (Jacket and Pants) and a control unit. The body Garments (Jacket and Pants) is a suit with 58 embedded electrodes that can stimulate 40 groups of muscles, conductive wires and connectors to a detachable control unit, whose intended purpose is to transmit electric pulses from the control unit to key nerves and corresponding muscle groups throughout the body. The control unit is a battery powered electrical device which sends low intensity electric pulses through connectors to the Body Garments which in turn transmits the pulses from the connectors to key nerves and corresponding muscle groups throughout the body.
  Arms: Active astimulation
Device: Exopulse Mollii suit (sham) — In the sham condition, the control unit will be programmed to start stimulating for 1 minute then it will shut off.
  Arms: Sham stimulation

SUMMARY:
Fibromyalgia is a debilitating pain condition that is characterized by the chronic occurrence of pain affecting the musculoskeletal system, a sensitivity to pressure stimuli, and a low threshold to noxious stimuli. The topography of pain is widespread, although it could be more pronounced in some bodily regions. Besides pain, patients suffer from a wide range of symptoms, including fatigue, anxiety and depression manifestations, and altered quality of life. Facing these debilitating symptoms, the available therapeutic strategies for treating pain and associated manifestations are usually faced with limited efficacy and numerous side effects. For these reasons, non-invasive stimulation techniques, namely transcutaneous stimulation by means of Exopulse Mollii suit, might be of help in this context.

The investigators designed a randomized sham controlled double-blind trial to demonstrate the improvement of pain, quality of life, fatigue and mood in adult patients with fibromyalgia following a 2-week intervention of "active" versus "sham" Exopulse Mollii suit. A 2-week washout period should be enough to prevent a potential carry over effect. After this phase (phase 1), a second open label phase (phase 2) will be proposed for patients to understand the effects of Exopulse Mollii suit employed for 4 weeks (7 sessions per week) on the studied outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years, with a definite diagnosis of fibromyalgia according to the American College of Rheumatology (ACR) 2010 criteria, set for at least one month
* Patients should be French speakers, able to understand verbal instructions, and affiliated to the national health insurance

Exclusion Criteria:

* Patient with VAS < 4
* Patient included in another research protocol during the study period
* Patient unable to undergo medical monitor for the study purposes due to geographical or social reasons
* Patient with contraindication to wearing Exopulse Mollii suit (e.g., cardiac stimulator, a ventriculoperitoneal shunt, intrathecal baclofen pump, pregnancy, and/or body mass index above 35 kg/m2)
* Patient with other somatic or psychiatric diagnoses other than anxiety and depression (e.g., arrhythmias, uncontrolled epilepsy, other diseases causing osteoarticular and muscular pain)
* Any change in the pharmacological therapy in the last three months
* Introduction of a medical device other than Exopulse Mollii suit during the study period
* Patient under juridical protection (" mesure de protection judiciare : tutelle, curatelle, sauvegarde de justice ")

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in the Visual Analogue Scale for Pain | This be assessed at baseline (before intervention) then at 2 weeks, 4 weeks, 6 weeks, 8 weeks and 12 weeks later
  VAS consists of rating the symptom on a 10 cm horizontal line going from "no pain" to "worst pain imaginable".

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS) | This be assessed at baseline (before intervention) then at 2 weeks, 4 weeks, 6 weeks, 8 weeks and 12 weeks later
  Pain Catastrophizing Scale (PCS) will be employed, which is a valid and reliable scale that includes 13 items assessing the presence and severity of feelings or thoughts that emerge when experiencing pain. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (all the time). It is possible to calculate a total and three subscale scores (i.e., helplessness, magnification, and rumination)
Brief Pain Inventory | This be assessed at baseline (before intervention) then at 2 weeks, 4 weeks, 6 weeks, 8 weeks and 12 weeks later
  The validated French version of the Brief Pain Inventory (BPI) will be used to assess pain severity (4 items) and pain interference (7 items). BPI items are rated on a 10-point scale running from 0 (no pain/does not interfere) to 10 (pain as bad as the participant can imagine/interferes completely).
Visual Analogue Scale (VAS) for fatigue | This be assessed at baseline (before intervention) then at 2 weeks, 4 weeks, 6 weeks, 8 weeks and 12 weeks later
  Like pain, fatigue will be assessed using VAS which consists of rating the symptom on a 10 cm horizontal line going from "no fatigue" to "worst fatigue imaginable".
Fibromyalgia Impact Questionnaire (FIQ) | This be assessed at baseline (before intervention) then at 2 weeks, 4 weeks, 6 weeks, 8 weeks and 12 weeks later
  It is an 11-item scale that assesses health status and functional disability by exploring the impact of fibromyalgia on work, wellbeing, fatigue, sleep, stiffness, anxiety, and depression. FIQ scores can range from 0 to 100, with higher scores reflecting worse health status. Scores could be used to classify fibromyalgia as mild (scores: 0-38), moderate (scores: 39-58), and severe (scores: 59-100)
Hospital Anxiety and Depression Scale (HADS) | This be assessed at baseline (before intervention) then at 2 weeks, 4 weeks, 6 weeks, 8 weeks and 12 weeks later
  It is a 14-item generic scale with good psychometric properties and consists of seven items assessing anxiety and seven others assessing depression. Scores can range from 0 to 21 on each subscale, with higher scores indicating worse symptomatology
Short Form 36 Health Survey (SF-36) | This be assessed at baseline (before intervention) then at 2 weeks, 4 weeks, 6 weeks, 8 weeks and 12 weeks later
  It is a generic survey that contains 36 items which assess the quality of life and yield eight dimensions: physical functioning, physical role, emotional role, bodily pain, general health, vitality, social functioning, and mental health. The score of each dimension ranges from 0 to 100, with higher scales implying better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Samar S. Ayache, MD, PhD, Principal Investigator — Clinical Neurophysiology department, Henri Mondor Hospital, Creteil, France
Locations (1):
- Hopital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No